CLINICAL TRIAL: NCT00740441
Title: A Phase II, Open Label, Single Arm Study of AS1411 in Patients With Metastatic Renal Cell Carcinoma
Brief Title: A Phase II Study of AS1411 in Renal Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Antisoma Research (Industry)
Responsible Party: Chris Smyth, Antisoma
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AS1411-C-202
Record Dates: First submitted 2008-08-22; First posted 2008-08-25 (Estimated); Last update posted 2009-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: renal cell carcinoma; rcc; kidney cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — AGRO 100

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): AS1411 treatment
  Interventions: Drug: AS1411

INTERVENTIONS:
Drug: AS1411 — AS1411 40 mg/kg/day) will be administered on days 1-4 via a continuous iv infusion every 28-day cycle for up to 2 cycles

SUMMARY:
The aim of this study is to evaluate the efficacy of AS1411 in patients with Metastatic Renal Cell Carcinoma

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed renal cell carcinoma containing predominant clear cell histology
* Failed or intolerant to 1 or more previous lines of treatments (which must include a Tyrosine Kinase Inhibitor)

Exclusion Criteria:

* Collecting duct histology
* A history of bleeding disorders or currently taking oral vitamin K antagonise medication
* Unstable brain metastases
* History of prior or concomitant malignancy (except for curatively treated non-melanoma skin cancer or carcinoma in situ of the cervix, or other cancer for which the patient has been disease free for 3 years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-09 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
To determine the Overall Response Rate to AS1411

SECONDARY OUTCOMES:
To measure progression free survival with AS1411
To measure time to disease progression with AS1411
To measure the duration of overall response and stable disease with AS1411
To determine the safety and tolerability of two cycles of AS1411
To assess the pharmacokinetic profile of AS1411
To assess pharmacodynamic markers of AS1411

CONTACTS AND LOCATIONS:
Overall Officials: Greg Smith, MD, Principal Investigator — Saint Francis Hospital; Harry Drabkin, MD, Principal Investigator — Medical University of South Carolina
Locations (7):
- United States (7):
  - City of Hope, Duarte, California
  - University of California, Davis Cancer Center, Sacramento, California
  - University of California San Francisco, San Francisco, California
  - St Francis Hospital, Beech Grove, Indiana
  - James Graham Brown Cancer Center, University of Louisville, Louisville, Kentucky
  - Lank Center for Genitourinary Oncology, Dana-Farber Cancer Institute, Boston, Massachusetts
  - Medical University of South Carolina, Charleston, South Carolina

REFERENCES:
- [Derived] Rosenberg JE, Bambury RM, Van Allen EM, Drabkin HA, Lara PN Jr, Harzstark AL, Wagle N, Figlin RA, Smith GW, Garraway LA, Choueiri T, Erlandsson F, Laber DA. A phase II trial of AS1411 (a novel nucleolin-targeted DNA aptamer) in metastatic renal cell carcinoma. Invest New Drugs. 2014 Feb;32(1):178-87. doi: 10.1007/s10637-013-0045-6. Epub 2013 Nov 16. PMID 24242861